CLINICAL TRIAL: NCT06912308
Title: Changes in Functional and Qualitative Indicators of Critically Ill Patients With Respiratory Failure Using Different Physiotherapy Methods
Brief Title: Effect of Physiotherapy Methods on Functional and Respiratory Outcomes in ICU Patients With Respiratory Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Rutkauskienė (Other)
Collaborators: Lithuanian University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Laura Rutkauskienė, Clinical Researcher, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Protocol number 1 • Version 3
Record Dates: First submitted 2025-03-16; First posted 2025-04-04 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Physiotherapy Intervention Arm (n=75) (Experimental): The subjects of one group will receive active physiotherapy (eg: verticalization, sitting on the edge of the bed, active breathing exercises).
  Interventions: Other: Active Physiotherapy
- Passive Physiotherapy Intervention Arm (n=75) (Experimental): The other group will receive passive physiotherapy methods (eg: passive movements, electrostimulation of the diaphragm).
  Interventions: Other: Passive Physiotherapy

INTERVENTIONS:
Other: Active Physiotherapy — Involves patient-driven exercises such as verticalization, sitting on the edge of the bed, and active breathing exercises.
  Arms: Active Physiotherapy Intervention Arm (n=75)
Other: Passive Physiotherapy — Employs methods like passive movements and electrostimulation of the diaphragm, providing therapeutic benefits without requiring active patient engagement.
  Arms: Passive Physiotherapy Intervention Arm (n=75)

SUMMARY:
The aim of the biomedical study is to assess the changes in functional and qualitative indicators of critically ill patients with respiratory failure by applying different physiotherapy methods. By conducting this study and developing the "Physiotherapy Protocol for Critically Ill Patients Treated in the ICU," physiotherapists worldwide could be encouraged to work using a unified and adapted method.

It is expected that the results, conclusions, and practical clinical recommendations derived from this study will be beneficial not only for rehabilitation specialists and intensivists in Lithuania but also for medical professionals working with respiratory diseases, including COVID-19 patients, at various stages of their treatment and consultation.

Implementing an appropriate physiotherapy procedure protocol is anticipated to bring economic benefits, as early physiotherapy is safe and can reduce the incidence of delirium, decrease the duration of patient sedation, shorten the number of days on mechanical ventilation, and minimize hospital stay duration. Additionally, it aims to restore or improve patients' functional and independence levels, help prevent ICU-acquired weakness, and can be easily implemented in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years of age)
* Hospitalized in the Department of Reanimation and Intensive Therapy at LSMU Kaunas Clinics
* Diagnosis of respiratory failure (KFN) based on the following TLK-10-AM codes: J96.00, J96.01, J96.9, J96.10, J96.11, J96.19, J96.90, J96.91, J96.99
* Signed informed consent obtained from the patient or their legal representative

Exclusion Criteria:

* Conscious patients who refuse to participate in the study
* Unconscious patients whose legal representative does not consent
* Recent episode of myocardial ischemia
* Pregnancy
* Heart rate < 40 bpm or > 130 bpm
* Mean arterial pressure < 60 mmHg or > 110 mmHg
* Oxygen saturation (SpO₂) ≤ 85%
* Body temperature ≥ 38.5°C or ≤ 36.0°C

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1) from baseline to ICU discharge | From Day 1 of ICU admission to ICU discharge (up to 50 days)
  Pulmonary function will be assessed using spirometry. The following parameters will be measured in liters and as percentages of predicted values: Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1). Measurements will be taken on Day 1 (baseline) and at ICU discharge. The mean change in FVC and FEV1 will be calculated to assess respiratory improvement.

SECONDARY OUTCOMES:
Change in Arterial Oxygenation Parameters (PaO₂, FiO₂, and PaO₂/FiO₂ Ratio) During ICU Stay | From Day 1 of ICU admission to ICU discharge (up to 50 days)
  Arterial blood gas analysis will be performed to monitor oxygenation. The following parameters will be recorded daily: arterial oxygen partial pressure (PaO₂, mmHg), inspired oxygen fraction (FiO₂), and their ratio (PaO₂/FiO₂). These values will be used to assess the progression of respiratory function and severity of respiratory failure. Mean changes from baseline to ICU discharge will be analyzed.
Change in Heart Rate and Arterial Blood Pressure Before and After Physiotherapy Session | Immediately before and immediately after each physiotherapy session, up to 50 days during ICU stay
  Heart rate (beats per minute) and arterial blood pressure (systolic and diastolic, mmHg) will be measured immediately before and after each physiotherapy session to evaluate acute cardiovascular responses. Data will be recorded daily throughout the ICU stay (up to 50 days). Mean changes will be analyzed.
Change in Intensive Care Unit Mobility Scale (ICUMS) Scores During ICU Stay | From Day 1 of physiotherapy to ICU discharge (up to 50 days)
  Patient mobility will be evaluated using the Intensive Care Unit Mobility Scale (ICUMS), which scores mobility from 0 (passive movements only) to 10 (independent ambulation). The scale will be administered at the beginning of each physiotherapy session. Mean score progression over time will be used to assess functional mobility changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No
For now, we do not have enough human and financial resources to share IPD, but if our circumstances change, we are open to reconsidering this decision.

REFERENCES:
- [Derived] Rutkauskiene L, Kubilius R, Tamosuitis T. Early mobilization, breathing exercises and chest wall oscillation in patients with bilateral pneumonia disease in the intensive care unit: a randomized clinical trial. BMC Pulm Med. 2025 Nov 25;26(1):20. doi: 10.1186/s12890-025-04028-7. PMID 41286729